CLINICAL TRIAL: NCT07308678
Title: Wound Closure in Venous Leg Ulcers (VLUs) Treated With AQUACEL® Ag+ Extra™ vs Cutimed® Sorbact®: A Blinded Re-Assessment of Randomized Controlled Trial Findings
Brief Title: AQUACEL® Ag+ Extra™ vs Cutimed® Sorbact®
Status: Completed | Type: Observational
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: WC-25-463
Record Dates: First submitted 2025-12-17; First posted 2025-12-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Venous Leg Ulcer; Diabetic Foot
MeSH Terms: conditions — Varicose Ulcer; Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study is to provide a blinded assessment of wound closure status utilizing photographs collected as per standard of care (SOC) during the AAA RCT (WC-22-435).

DETAILED DESCRIPTION:
The purpose of the study is to provide a blinded (treatment arm, timepoint) assessment of wound closure status utilizing photographs collected as per standard of care (SOC) during the AAA Randomized Controlled Trial (RCT) (WC-22-435).

ELIGIBILITY:
Inclusion Criteria:

* All subjects from the intention to treat (ITT) population with wound photograph(s) corresponding to the study visit date (WC-22-435) indicating wound closure or their 12-week visit, whichever came first

Exclusion Criteria:

* Subjects whose photographs are deemed of insufficient quality to make determination of closure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have wound photographs of sufficient quality taken as per standard of care (SOC) during the AAA RCT (WC-22-435) that correspond to wound closure or their 12-week visit.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Wound closure at 12 weeks | 12 week
  Incidence of wound closure at 12 weeks, defined as 100% epithelialization of the wound surface, assessed by a blinded observer through photographic evidence

OTHER OUTCOMES:
Inter-rater reliability of photographic assessment | up to 12 week
  Inter-rater reliability (IRR) of photographic to live assessment of wound closure
Inter-rater reliability of photographic site assessment | up to 12 week
  IRR of photographic to live assessment of wound closure, by study site

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Dissemond, MD, Principal Investigator — Essen University Hospital
Locations (1):
- Essen University Hospital, Essen, Germany